CLINICAL TRIAL: NCT01811316
Title: A Clinical Trial to Evaluate Long-term Efficacy and Safety of Lozenges Containing Lactobacilli Reuteri (Prodentis™) on Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLP-2013-1-23
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotics Lozenge (twice a day) (Active Comparator): Subjects take their lozenge twice a day, one lozenge in the morning after brushing and one lozenge in the evening after brushing.
  Interventions: Other: Probiotics
- Probiotics Lozenge (once a day) (Active Comparator): Subjects take their lozenge once a day, one lozenge at night after brushing.
  Interventions: Other: Probiotics
- Placebo Lozenge (once a day) (Placebo Comparator): Subjects take their lozenge once a day, one lozenge at night after brushing.
  Interventions: Other: Probiotics

INTERVENTIONS:
Other: Probiotics

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of lozenges containing probiotics in reducing gingivitis. The primary purpose of this study is to support claims from U.S. instructions for use (IFU) for GUM® PerioBalance®.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, understand and sign an Informed Consent form.
* Good general health as evidenced by the medical history.
* Between 18 and 65 years of age.
* Male or female.
* Minimum of 20 teeth, excluding crowns and third molar teeth.
* Mean whole mouth Modified Gingival Index of greater-than or equal to 2.0 at baseline.
* Willing to abstain from all oral hygiene procedures for 12-18 hours prior to clinical visits.
* Willing to abstain from eating and drinking in the morning of visits, only drinking water is allowed.
* Willing to abstain from interdental cleaning, chewing gums, oral whitening, mouth rinse and tobacco products for the study duration.
* Able to understand and follow study directions.
* No known history of allergy to dairy products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria

* Presence of orthodontic appliances.
* Intra-oral soft tissue lesions due to pathology or trauma
* Patients with aggressive periodontitis, acute necrotizing ulcerative gingivitis, or gross decay at discretion of PI.
* More than two sites with pocket depth >5mm and concomitant attachment loss of >2mm.
* Pregnant or lactating females or females of child bearing potential not using acceptable methods of birth control (hormonal, barriers or abstinence).
* Use of antibiotics within 3 months of enrollment
* History of drug use that is associated with gum overgrowth (i.e., Dilantin, nifedipine, etc)
* Chronic use of medication such as steroids, NSAIDs (more than 2-3 days/week), anti-coagulant medications, immunosuppressant medications or any other medications that in the opinion of the Investigator would interfere with the evaluation or confound interpretation of the study results. Use of low dose of acetylsalicylic acid (81 mg) is permitted.
* Unwilling to sign a confidentiality statement and/or return the test products.
* Medical condition which requires pre-medication prior to dental visits/procedures.
* Immune compromised individuals (HIV, AIDS, immunosuppressive drug therapy).
* Current use of probiotics or probiotic containing food (i.e., yogurt)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hasturk, DDS, PhD, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Started | 21 | 22 | 19
Visit 4 Weeks | 19 | 22 | 19
Visit 12 Weeks | 18 | 22 | 19
Completed | 18 | 22 | 19
Not Completed | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day) | Total
Number analyzed (Participants) | 21 | 22 | 19 | 62
Age, Continuous [Mean (Standard Deviation); unit: Year] | 40 (13) | 44 (15) | 34 (11) | 40 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 9 | 32
  Male | 11 | 9 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 19 | 21 | 19 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 7 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 5 | 1 | 4 | 10
  White | 12 | 12 | 10 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Gingival Index (MGI)
Description: Modified Gingival Index (MGI) (Lobene, Weatherford et al. 1986) was measured on six gingival areas of all scorable teeth, using a scale of 0-4 as follows: Scores Criteria 0 Normal (absence of inflammation)
  1. Mild inflammation (slight change of color, little change in texture) of any portion of, but not the entire marginal or papillary gingival unit
  2. Mild inflammation of the entire gingival unit
  3. Moderate inflammation (moderate glazing, redness, edema and/or hypertrophy) of the marginal or papillary gingival unit
  4. Severe inflammation (marked redness and edema/hyper-trophy, spontaneous bleeding or ulceration) of the marginal or papillary gingival unit.
  Whole mouth MGI scores were calculated by summing all scores and dividing by the number of examined scorable sites.
Time Frame: 4, 12 and 24 weeks
Population: One subject was lost to follow up between 4 and 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Number analyzed (Participants) | 19 | 22 | 18
units on a scale
  4 weeks | -0.07 (0.12) | -0.09 (0.12) | -0.09 (0.12)
  12 weeks: number analyzed (Participants) | 18 | 22 | 18
  12 weeks | -0.02 (0.11) | -0.02 (0.12) | -0.04 (0.11)
  24 weeks: number analyzed (Participants) | 18 | 22 | 18
  24 weeks | 0.00 (0.13) | -0.04 (0.13) | -0.06 (0.12)

2. Primary Outcome: Change From Baseline in Bleeding on Probing (BOP)
Description: Bleeding on probing was assessed 30 seconds after probing. A dichotomous scoring system was used at six sites per tooth using one (1) and zero (0) for presence or absence, respectively. BOP (%) is a percentage of sites BOP.
Time Frame: 4, 12 and 24 weeks
Population: One subject was lost to follow up between 4 and 12 weeks.
Measure: Mean (Standard Deviation); unit: percentage of sites BOP
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Number analyzed (Participants) | 19 | 22 | 19
percentage of sites BOP
  4 weeks | -10.2 (13.8) | -1.8 (10.7) | -3.0 (9.2)
  12 weeks: number analyzed (Participants) | 18 | 22 | 19
  12 weeks | -6.6 (14.9) | 0.8 (13.5) | 2.9 (14.5)
  24 weeks: number analyzed (Participants) | 18 | 22 | 19
  24 weeks | -2.3 (17.1) | 5.6 (17.9) | 3.5 (14.1)

3. Secondary Outcome: Change From Baseline in Plaque Index (PI)
Description: Plaque Index of Turesky Modification of Quigley-Hein (Turesky, Gilmore et al. 1970) (PI) was scored on all natural teeth (except third molars) after disclosing with erythrosine solution. Scores Criteria:
  0 No plaque
  1. Separate flecks of plaque at the cervical margin of the tooth
  2. A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth
  3. A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  4. Plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. Plaque covering two-thirds or more of the crown of the tooth
Time Frame: 4, 12 and 24 weeks
Population: One subject was lost to follow up between 4 and 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Number analyzed (Participants) | 19 | 22 | 18
units on a scale
  4 weeks | 0.08 (0.36) | 0.06 (0.28) | 0.08 (0.49)
  12 weeks: number analyzed (Participants) | 18 | 22 | 18
  12 weeks | 0.18 (0.35) | 0.06 (0.4) | 0.00 (0.54)
  24 weeks: number analyzed (Participants) | 18 | 22 | 18
  24 weeks | 0.25 (0.44) | 0.11 (0.39) | 0.03 (0.47)

4. Secondary Outcome: Change From Baseline in Probing Depth (PD)
Description: Periodontal pocket depth (PD) was determined with a periodontal probe at six sites per tooth rounded to the next lower whole mm.
Time Frame: 4, 12 and 24 weeks
Population: One subject was lost to follow up between 4 and 12 weeks.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Number analyzed (Participants) | 19 | 22 | 19
mm
  4 weeks | 0.01 (0.11) | 0.00 (0.13) | 0.02 (0.13)
  12 weeks: number analyzed (Participants) | 18 | 22 | 19
  12 weeks | 0.01 (0.12) | 0.03 (0.12) | 0.10 (0.15)
  24 weeks: number analyzed (Participants) | 18 | 22 | 19
  24 weeks | 0.1 (0.11) | 0.08 (0.15) | 0.11 (0.19)

5. Other Pre Specified Outcome: Change From Baseline in Inflammatory Markers in Gingival Crevicular
Description: Gingival Crevicular Fluid (GCF) samples will be analyzed for inflammatory cytokines/chemokines and matrix metalloproteases using multiplexing ELISA.
Time Frame: 15 days, 4, 12 and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected at each visit over 24 weeks after randomization.
Arm/Group | Probiotics Lozenge (Twice a Day) | Probiotics Lozenge (Once a Day) | Placebo Lozenge (Once a Day)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 1/21 | 2/22 | 5/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotics Lozenge (Twice a Day) (N=21) | Probiotics Lozenge (Once a Day) (N=22) | Placebo Lozenge (Once a Day) (N=19)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sore throat (Social circumstances) | 1 (1) | 0 (0) | 1 (1)
Allergic sinustis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. PI shall delay publications for up to 90 days upon receipt of a written request from the sponsor in order to allow the sponsor to register intellectual property rights that are included in the proposed publication.